CLINICAL TRIAL: NCT03523182
Title: Promoting Spirulina Production and Utilization in Luapula Province of Zambia
Brief Title: Spirulina Supplementation and Infant Growth, Morbidity and Motor Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Programme Against Malnutrition (Other)
Collaborators: Hitotsubashi University (Other); Alliance Forum Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FWA00000338
Record Dates: First submitted 2018-04-19; First posted 2018-05-14 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Stunting; Underweight; Pneumonia, Pneumocystis; Cough; Malaria; Fever; Motor Delay
Keywords: Micronutrient supplementation; Home fortification; Spirulina; Zambia
MeSH Terms: conditions — Growth Disorders; Thinness; Pneumonia, Pneumocystis; Cough; Malaria; Fever; Psychomotor Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spirulina (SP) (Experimental): Children in the SP group (n=251) received a soya-maize-based porridge for 12 months with the addition of spirulina.
  Interventions: Dietary Supplement: Spirulina; Dietary Supplement: Control
- Control (CON) (Active Comparator): Children in the CON group (n=250) received a soya-maize-based porridge for 12 months.
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Spirulina — Arthrospira platensis, also known as spirulina, is a blue-green micro-algae indigenous to Africa.
  Spirulina group (n=251) receive a soya-maize-based porridge with the addition of spirulina.
  We used 10 g per day of spirulina powder with a mealie meal and soya flour porridge blend.
  Arms: Spirulina (SP)
Dietary Supplement: Control — Children receive a soya-maize-based porridge for 12 months. We use a mealie meal and soya flour porridge blend.

SUMMARY:
Background: In developing countries, micronutrient deficiency in infants is associated with growth faltering, morbidity, and delayed motor development. One of the potentially low-cost and sustainable solutions is to use locally producible food for the home fortification of complementary foods.

Objective: The objectives are to test the hypothesis that locally producible spirulina platensis supplementation would achieve the following: 1) increase infant physical growth; 2) reduce morbidity; and 3) improve motor development.

Design: 501 Zambian infants are randomly assigned into a control (CON) group or a spirulina (SP) group. Children in the CON group (n=250) receive a soya-maize-based porridge for 12 months, whereas those in the SP group (n=251) receive the same food but with the addition of spirulina. The change in infants' anthropometric status, morbidity, and motor development over 12 months are assessed.

DETAILED DESCRIPTION:
Micronutrient deficiency in the infancy is associated with growth faltering, morbidity, and delayed motor development, and is common in developing countries where the food available for infants has low micronutrient density.

A low-cost and sustainable way to address this problem is to utilize locally producible foods rich in multi-micronutrients as home supplements to complementary food. Arthrospira platensis, also known as spirulina, is a blue-green micro-algae indigenous to Africa.

It contains a high percentage of protein, and is rich in multiple micronutrients know to support infant growth such as beta carotene, B vitamins, and minerals such as calcium, iron, magnesium, manganese, potassium, and zinc. The cost of producing spirulina is much lower than that of producing other comparably protein-rich foods, such as soya beans and beef, and therefore may potentially sustainably meet the nutritional demands of African infants.

Our objective is to assess the acceptability and effects of spirulina supplementation on growth, incidence of morbidity, and level of motor development in infants in Zambia. The testable hypothesis is that spirulina supplementation for 12 months would increase infant height, reduce the incidence of morbidity, and reduce time taken to achieve motor development milestones (ability to walk unassisted).

This study is conducted from April 2015 to April 2016 in the form of an open-labeled randomized control trial, and involves in a spirulina-fed treatment (SP) group and a control (CON) group.

501 Zambian infants are randomly assigned into a control (CON) group or a spirulina (SP) group. Children in the CON group (n=250) receive a soya-maize-based porridge for 12 months, whereas those in the SP group (n=251) receive the same food but with the addition of spirulina.

The change in infants' anthropometric status, morbidity, and motor development over 12 months are assessed.

Amendment: the study period has been extended by 4 months. Without no-intervention period, monthly supplementation was restarted in study are.

ELIGIBILITY:
Inclusion Criteria:

* All infants were eligible for the study if they are between 6 and 18 month of age

Exclusion Criteria:

* Non-singleton birth infants were excluded

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 501 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in height-for-age z-scores (HAZ) at 32 month follow up | Height of the infants are measured by experienced field workers at at 0, 6, and 12 month. Amendment: also measured at extension endline (October 2016), at 24 month follow up (April 2017) and at 32 month follow up (January 2018) survey.
  Primary outcome is changes in HAZ. Height of the infants is transformed to standardized scores using the World Health Organization (WHO) Multicentre Growth Standards
Child development | At 32 month follow up (January 2018) survey
  Study children will be assessed at 32 month follow up (January 2018) using the Malawi Development Assessment Tool (MDAT) instrument. Scores will be standardized within the study sample for analysis. Scores of children in treatment group will be compared with children in comparison group to determine differences.

SECONDARY OUTCOMES:
Change from baseline in weight-for-age z-scores (WAZ) at 32 month follow up | Weight of the infants are measured at 0, 6, and 12 month by experienced field workers. Amendment: also measured at extension endline (October 2016), at 24 month follow up (April 2017) and at 32 month follow up (January 2018)
  Secondary outcome is changes in WAZ. Weight of the infants is transformed to standardized scores using the WHO Multicentre Growth Standards
Change from baseline in pneumonia incidence at 32 month follow up | Data on pneumonia indicators were collected up to 12 months by trained local health workers. Amendment: also measured at extension endline (October 2016), at 24 month follow up (April 2017) and at 32 month follow up (January 2018)
  Secondary outcome is changes in pneumonia incidence. Pneumonia was defined as cough accompanied by short and rapid breathing and difficulty in breathing
Change from baseline in cough incidence at 32 month follow up | Data on cough morbidity indicators are collected up to 12 months by trained local health workers. Amendment: also measured at extension endline (October 2016), at 24 month follow up (April 2017) and at 32 month follow up (January 2018)
  Secondary outcome is changes in cough incidence in the 4 weeks preceding the interview.
Change from baseline in severe high fever incidence at 32 month follow up | Data are collected up to 12 months by trained local health workers. Amendment: also measured at extension endline (October 2016), at 24 month follow up (April 2017) and at 32 month follow up (January 2018)
  Secondary outcome is changes in severe high fever incidence. Severe high fever was defined based on the following clinical signs: fever with rash on child's body, fever with chills, shaking, nausea, or alternating high and low body temperature
Change from baseline in fever incidence at 32 month follow up | Data are collected up to 12 months by trained local health workers. Amendment: also measured at extension endline (October 2016), at 24 month follow up (April 2017) and at 32 month follow up (January 2018)
  Secondary outcome is changes in fever incidence in the 4 weeks preceding the interview
Ability of the infant to walk independently. | This indicator was evaluated at 0, 6 and 12 months by research assistants who visited the participants' homes
  The ability of children to walk without assistance measured by the questionnaire.
Child development at 24 month follow up | At 24 month follow up survey (April 2017)
  Study children will be assessed at 24 month follow up (April 2017) using the Malawi Development Assessment Tool (MDAT) instrument. Scores will be standardized within the study sample for analysis. Scores of children in treatment group will be compared with children in comparison group to determine differences.

CONTACTS AND LOCATIONS:
Overall Officials: Kazuya Masuda, PhD, Principal Investigator — Hitotsubashi University
Locations (1):
- Programme Against Malnutrition, Mansa, Luapura, Zambia

IPD SHARING:
Plan to Share IPD: No